CLINICAL TRIAL: NCT00697515
Title: A Phase IIIb Randomized, Double-Blind, Multicenter, Placebo-Controlled, Dose Optimization, Crossover, Safety and Efficacy Workplace Environment Study of Lisdexamfetamine Dimesylate (LDX) in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Brief Title: Safety and Efficacy Workplace Environment Study of Lisdexamfetamine Dimesylate (LDX) in Adults With Attention-Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SPD489-316
Record Dates: First submitted 2008-06-11; First posted 2008-06-16 (Estimated); Results first posted 2010-02-01 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine Dimesylate (LDX, SPD489) (Active Comparator)
  Interventions: Drug: LDX
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LDX — oral, 30, 50, or 70 mg once-daily for 4 weeks during dose optimization, and then for 1 week during each crossover during the adult workplace environment setting
  Arms: Lisdexamfetamine Dimesylate (LDX, SPD489)
Drug: Placebo — Placebo administered once-daily for one week during the adult workplace environment setting
  Arms: Placebo

SUMMARY:
To evaluate the efficacy of LDX compared to placebo in adults with ADHD in the adult workplace environment (AWE) setting

DETAILED DESCRIPTION:
This study has both an optimization and double-blind period

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18-55 years of age, inclusive at the time of consent.
* Female subjects must have a negative serum beta Human Chorionic Gonadotropin (HCG) pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to comply with any applicable contraceptive requirements of the protocol.
* Subject meets Diagnostic and Statistical Manual of Mental Disorders Fourth Edition; Text Revision (DSM IV TR) criteria for a primary diagnosis of ADHD (diagnostic code 314.00 and 314.01) established by a comprehensive psychiatric evaluation that reviews DSM-IV-TR criteria with at least 6 of the 9 subtype criteria met. The Adult ADHD Clinical Diagnostic Scale version 1.2 (ACDS v1.2) will be utilized as the diagnostic tool.
* Subject has a Baseline score of > or equal to 28 using the Adult ADHD-RS with prompts.
* Subject must have a minimum level of intellectual functioning, as determined by an Intelligent Quotient (IQ) score of 80 or above based on the Kaufman Brief Intelligence Test (KBIT).

Exclusion Criteria:

* Subject has a current comorbid psychiatric disorder that is either controlled with medications prohibited in this study or is uncontrolled and associated with significant symptoms. Comorbid psychiatric diagnoses will be established by the psychiatric evaluation that includes the Structured Clinical Interview for DSM-IV-TR disorders (SCID-I).
* Subjects who are currently considered a suicide risk, any subject who has previously made a suicide attempt or those who are currently demonstrating active suicidal ideation.
* Subject has a history of seizures (other than infantile febrile seizures), any tic disorder, or a current diagnosis and/or a known family history of Tourette's Disorder.
* Subject has known history of symptomatic cardiovascular disease, advanced arteriosclerosis, structural cardiac abnormality, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, transient ischemic attack or stroke or other serious cardiac problems that may place them at increased vulnerability to the sympathomimetic effects of a stimulant drug.
* Subject has current abnormal thyroid function, as defined as abnormal Screening thyroid stimulating hormone. Treatment with a stable dose of thyroid medication for at least 3 months is permitted.
* Subject has a history of moderate to severe hypertension or has a resting sitting systolic blood pressure >139mmHg or diastolic blood pressure >89mmHg.
* Subject has a documented allergy, hypersensitivity, or intolerance to amphetamines.
* Subject has failed to respond to one or more adequate courses (dose and duration) of amphetamine therapy.
* Subject has glaucoma.
* Subject is taking other medications that have central nervous system (CNS) effects or affect performance, such as sedating antihistamines and decongestant sympathomimetics, or are monoamine oxidase inhibitors (during or within 14 days of test or reference product administration). Stable use of bronchodilator inhalers is not exclusionary.
* Subject is female and pregnant or lactating.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2008-07-18 (Actual); Primary Completion 2008-12-20 (Actual); Study Completion 2008-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Clinical Study Centers, LLC, Little Rock, Arkansas
  - University of CA, Irvine Child Development Center, Irvine, California
  - Vince & Associates Clinical Research, Overland Park, Kansas
  - Center for Psychiatry & Behavioral Medicine, Inc, Las Vegas, Nevada
  - Bayou City Research, LTD, Houston, Texas

REFERENCES:
- [Result] Wigal T, Brams M, Gasior M, Gao J, Squires L, Giblin J; 316 Study Group. Randomized, double-blind, placebo-controlled, crossover study of the efficacy and safety of lisdexamfetamine dimesylate in adults with attention-deficit/hyperactivity disorder: novel findings using a simulated adult workplace environment design. Behav Brain Funct. 2010 Jun 24;6:34. doi: 10.1186/1744-9081-6-34. PMID 20576091
- [Result] Brams M, Giblin J, Gasior M, Gao J, Wigal T. Effects of open-label lisdexamfetamine dimesylate on self-reported quality of life in adults with ADHD. Postgrad Med. 2011 May;123(3):99-108. doi: 10.3810/pgm.2011.05.2288. PMID 21566420
- [Result] Brown TE, Brams M, Gasior M, Adeyi B, Babcock T, Dirks B, Scheckner B, Wigal T. Clinical utility of ADHD symptom thresholds to assess normalization of executive function with lisdexamfetamine dimesylate treatment in adults. Curr Med Res Opin. 2011;27 Suppl 2:23-33. doi: 10.1185/03007995.2011.605441. PMID 21973229
- [Derived] Brown TE, Brams M, Gao J, Gasior M, Childress A. Open-label administration of lisdexamfetamine dimesylate improves executive function impairments and symptoms of attention-deficit/hyperactivity disorder in adults. Postgrad Med. 2010 Sep;122(5):7-17. doi: 10.3810/pgm.2010.09.2196. PMID 20861583
- See also: FDA recall information — http://www.fda.gov/opacom/7alerts.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study consisted of a 4-week dose optimization phase (30, 50 or 70 mg SPD489 once-daily) and a 2-week crossover phase. Of the 142 subjects enrolled in the dose optimization phase, 15 discontinued prior to randomization.
Groups:
- SPD489 First: Lisdexamfetamine Dimesylate (LDX, SPD489) is dosed once-daily at 30, 50 or 70 mg for 1 week during the first intervention and placebo is administered once-daily for 1 week in the second intervention.
- Placebo First: Placebo is administered once-daily for 1 week in the first intervention and Lisdexamfetamine Dimesylate (LDX, SPD489)is dosed once-daily at 30, 50 or 70 mg for 1 week during the second intervention.
Period: Dose Optimization Period
Arm/Group | SPD489 First | Placebo First
Started | 142 | 0
Completed | 127 | 0
Not Completed | 15 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — sponsor request | 2 | 0
Not completed — called to active duty | 1 | 0
Not completed — elevated QTc | 1 | 0
Period: First Intervention (Crossover Period)
Arm/Group | SPD489 First | Placebo First
Started | 63 | 64
Completed | 53 | 52
Not Completed | 10 | 12
Not completed — Natural disaster | 8 | 9
Not completed — Adverse Event | 0 | 2
Not completed — Withdrawal by Subject | 2 | 1
Period: Second Intervention (Crossover Period)
Arm/Group | SPD489 First | Placebo First
Started | 53 | 52
Completed | 52 | 51
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 142
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 142
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54
  Male | 88
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 142

OUTCOME MEASURES:

1. Primary Outcome: Permanent Product Measure of Performance (PERMP) Total Score Over the Treatment Day in the Crossover Phase
Description: The Permanent Product Measure of Performance (PERMP) is a skill adjusted math test. The PERMP score is the sum of the number of math problems attempted plus the number of math problems answered correctly in a 10-minute session. The scores range from 0-800 with higher scores indicating better performance.
Time Frame: 2, 4, 8, 10, 12 and 14 hours post-dose on Day 7
Population: Intent to Treat (ITT) population defined as all subjects who are randomized and have at least one post-dose primary efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- SPD489: Lisdexamfetamine Dimesylate (LDX, SPD489) is dosed once-daily at 30, 50 or 70 mg
- Placebo: Placebo is administered once-daily
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 104 | 104
Units on a scale | 312.9 (8.59) | 289.5 (8.59)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

2. Secondary Outcome: PERMP Total Score by Timepoint in the Crossover Phase
Description: as for outcome 1
Time Frame: 2, 4, 8, 10, 12 and 14 hours post-dose on Day 7
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 104 | 104
Units on a scale
  2.0 hours post-dose | 301.5 (8.78) | 285.9 (8.78)
  4.0 hours post-dose | 314.1 (9.16) | 284.7 (9.16)
  8.0 hours post-dose | 311.4 (9.07) | 287.1 (9.07)
  10.0 hours post-dose | 313.5 (8.82) | 288.8 (8.82)
  12.0 hours post-dose | 318.7 (8.77) | 293.1 (8.77)
  14.0 hours post-dose | 318.6 (9.03) | 296.7 (9.03)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; 2.0 hours post-dose; Test type: Superiority or Other; p = 0.0017, ANOVA
Statistical Analysis 2: Comparison: SPD489 vs Placebo; 4.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 3: Comparison: SPD489 vs Placebo; 8.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: SPD489 vs Placebo; 10.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: SPD489 vs Placebo; 12.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: SPD489 vs Placebo; 14.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA

3. Secondary Outcome: PERMP Score for the Number of Math Problems Attempted by Timepoint in the Crossover Phase
Description: as for outcome 1
Time Frame: 2, 4, 8, 10, 12 and 14 hours post-dose on Day 7
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 104 | 104
Units on a scale
  Over the treatment day | 158.6 (4.33) | 146.6 (4.33)
  2.0 hours post-dose | 153.1 (4.41) | 144.9 (4.41)
  4.0 hours post-dose | 159.3 (4.60) | 144.2 (4.60)
  8.0 hours post-dose | 157.6 (4.56) | 145.3 (4.56)
  10.0 hours post-dose | 158.6 (4.44) | 146.1 (4.44)
  12.0 hours post-dose | 161.2 (4.43) | 148.4 (4.43)
  14.0 hours post-dose | 161.5 (4.57) | 150.4 (4.57)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Average over the treatment day; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: SPD489 vs Placebo; 2.0 hours post-dose; Test type: Superiority or Other; p = 0.0010, ANOVA
Statistical Analysis 3: Comparison: SPD489 vs Placebo; 4.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: SPD489 vs Placebo; 8.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: SPD489 vs Placebo; 10.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: SPD489 vs Placebo; 12.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: SPD489 vs Placebo; 14.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA

4. Secondary Outcome: PERMP Score for the Number of Math Problems Answered Correctly by Timepoint in the Crossover Phase
Description: as for outcome 1
Time Frame: 2, 4, 8, 10, 12 and 14 hours post-dose on Day 7
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 104 | 104
Units on a scale
  Over the treatment day | 154.4 (4.27) | 142.9 (4.27)
  2.0 hours post-dose | 148.4 (4.38) | 141.0 (4.38)
  4.0 hours post-dose | 154.8 (4.56) | 140.4 (4.56)
  8.0 hours post-dose | 153.7 (4.51) | 141.7 (4.51)
  10.0 hours post-dose | 154.8 (4.39) | 142.7 (4.39)
  12.0 hours post-dose | 157.4 (4.36) | 144.7 (4.36)
  14.0 hours post-dose | 157.1 (4.48) | 146.3 (4.48)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Over the treatment day; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: SPD489 vs Placebo; 2.0 hours post-dose; Test type: Superiority or Other; p = 0.0031, ANOVA
Statistical Analysis 3: Comparison: SPD489 vs Placebo; 4.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: SPD489 vs Placebo; 8.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 5: Comparison: SPD489 vs Placebo; 10.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 6: Comparison: SPD489 vs Placebo; 12.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 7: Comparison: SPD489 vs Placebo; 14.0 hours post-dose; Test type: Superiority or Other; p < 0.0001, ANOVA

5. Secondary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale With Prompts (ADHD-RS) Total Score at up to 28 Days in the Dose Optimization Phase
Description: The Attention Deficit Hyperactivity Disorder Rating Scale with Prompts (ADHD-RS) consists of 18 items scored on a 4-point scale ranging from 0 (no symptoms) to 3 (severe symptoms) with total score ranging from 0 to 54.
Time Frame: Baseline and 7, 14, 21 and 28 days
Population: Enrolled Efficacy Population (EEP) defined as all subjects who have taken one dose of study medication in the Dose Optimization Phase and had one post-Baseline efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 142
Units on a scale | -21.4 (7.31)
Statistical Analysis 1: Comparison: SPD489; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

6. Secondary Outcome: ADHD-RS With Prompts Total Score in the Crossover Phase
Description: as for outcome 5
Time Frame: 7 days
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 104 | 104
Units on a scale | 18.1 (0.94) | 29.6 (0.94)
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, ANOVA

7. Secondary Outcome: Assessment of Clinical Global Impression-Severity of Illness (CGI-S) in the Dose Optimization Phase
Description: CGI-S assesses the severity of the subject's condition on a 7-point scale ranging from 1 (normal, not at all ill) to 7 (among the most extremely ill)
Time Frame: Baseline
Population: EEP
Measure: Number; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 142
Participants
  Normal, not at all ill | 0
  Borderline mentally ill | 0
  Mildly ill | 0
  Moderately ill | 92
  Markedly ill | 46
  Severely ill | 4
  Among the most extremely ill subjects | 0

8. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) in the Dose Optimization Phase
Description: CGI-I consists of a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Improvement is defined as a score of 1 (very much improved) or 2 (much improved) on the scale.
Time Frame: 7, 14, 21 and 28 days
Population: EEP
Measure: Number; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 132
Participants | 130

9. Secondary Outcome: Number of Participants With Improvement on Clinical Global Impression-Improvement (CGI-I) in the Crossover Phase
Description: as for outcome 8
Time Frame: 7 days
Population: ITT
Measure: Number; unit: Participants
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 103 | 103
Participants | 70 | 13
Statistical Analysis 1: Comparison: SPD489 vs Placebo; Test type: Superiority or Other; p < 0.0001, Prescott's Test

10. Secondary Outcome: Change From Baseline in the Brown Attention Deficit Disorder Scale (BADDS) Total Scores at 26 Days in the Dose Optimization Phase
Description: The BADDS assessment consists of 40 items rated on a scale from 0 (never) to 3 (almost daily). The total score ranges from 0 to 120 with increasing scores indicating more severe impairment.
Time Frame: Baseline and 26 days
Population: EEP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 127
Units on a scale | -34.1 (20.99)
Statistical Analysis 1: Comparison: SPD489; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

11. Secondary Outcome: Level of Satisfaction With Study Treatment on Medication Satisfaction Questionnaire (MSQ) in the Dose Optimization Phase
Description: MSQ is a survey rating the subject's level of satisfaction with the study treatment medication.
Time Frame: 26 days
Population: EEP
Measure: Number; unit: Participants
Arm/Group | SPD489
Number analyzed (Participants) | 127
Participants
  Very satisfied | 79
  Moderately satisfied | 44
  Not satisfied | 2
  Don't know | 2

12. Secondary Outcome: Change From Baseline in Adult ADHD Impact Module (AIM-A) Question 1 Score at 26 Days in the Dose Optimization Phase
Description: AIM-A is a quality of life instrument. Question 1 is 'On a scale of 1 to 10, how would you rate the overall quality of life right now?' It is rated on a scale of 1 (worst) to 10 (best).
Time Frame: Baseline and 26 days
Population: EEP
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 127
Units on a scale | 0.9 (1.67)
Statistical Analysis 1: Comparison: SPD489; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

13. Secondary Outcome: Change From Baseline in AIM-A Question 4 Score at 26 Days in the Dose Optimization Phase
Description: AIM-A is a quality of life instrument. Question 4 is 'How much do you agree with this statement: Over the past few weeks, I've had more good days than bad days?' This is rated on a scale of 1 (strongly agree) to 5 (strongly disagree).
Time Frame: Baseline and 26 days
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | SPD489
Number analyzed (Participants) | 127
Units on a scale | -0.7 (0.96)
Statistical Analysis 1: Comparison: SPD489; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure at Up to 28 Days in the Dose Optimization Phase
Time Frame: Baseline and 7, 14, 21 and 28 days
Population: Safety Population (SP) defined as all subjects who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SPD489
Number analyzed (Participants) | 142
mmHg | -0.3 (9.46)

15. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure at Up to 28 Days in the Dose Optimization Phase
Time Frame: Baseline and 7, 14, 21 and 28 days
Population: SP
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | SPD489
Number analyzed (Participants) | 142
mmHg | -0.2 (6.94)

16. Secondary Outcome: Change From Baseline in Pulse Rate at Up to 28 Days in the Dose Optimization Phase
Time Frame: Baseline and 7, 14, 21 and 28 days
Population: SP
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | SPD489
Number analyzed (Participants) | 142
bpm | 3.2 (11.55)

17. Secondary Outcome: Change From Baseline in Electrocardiogram Results (QTcF Interval) at 7 Days in the Crossover Phase
Description: QTcF is the QT interval using Fridericia's correction formula. QT interval is a measure of time between the start of the Q wave and the end of the T wave and is dependent on the heart rate(e.g., the faster the heart rate, the shorter the QT interval). The QT interval has to be corrected in order to aid interpretation.
Time Frame: Baseline and 7 days
Population: SP
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | SPD489 | Placebo
Number analyzed (Participants) | 115 | 117
msec | 4.4 (16.62) | 4.8 (15.45)

ADVERSE EVENTS:
Description: Safety Population defined as all subjects who received at least one dose of study medication. All 142 subjects received at least one dose of study medication during the dose optimization phase. In the crossover phase, 64 subjects received placebo in the first intervention and 53 in the second intervention for a total of 117 for placebo.
Groups:
- SPD489: Lisdexamfetamine Dimesylate (LDX, SPD489) is dosed once-daily at 30, 50 or 70 mg for 1 week during the first intervention and placebo is administered once-daily for 1 week in the second intervention.
- Placebo: Placebo is administered once-daily for 1 week in the first intervention and Lisdexamfetamine Dimesylate (LDX, SPD489)is dosed once-daily at 30, 50 or 70 mg for 1 week during the second intervention.
Arm/Group | SPD489 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/117
Other Adverse Events (participants affected / at risk) | 113/142 | 23/117
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SPD489 (N=142) | Placebo (N=117)
Dry mouth (Gastrointestinal disorders) | 43 | 0
Nausea (Gastrointestinal disorders) | 11 | 0
Feeling jittery (General disorders) | 8 | 0
Irritability (General disorders) | 12 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 9
Decreased appetite (Metabolism and nutrition disorders) | 52 | 0
Headache (Nervous system disorders) | 28 | 0
Anxiety (Psychiatric disorders) | 8 | 0
Insomnia (Psychiatric disorders) | 26 | 0
Fatigue (General disorders) | 0 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.